CLINICAL TRIAL: NCT05780294
Title: A Multi-center, Randomized, Double-blind, Phase III Clinical Trial of Leucogen Versus Placebo on Leukocyte and Platelet Whole-course Management Assisted by Platinum Plus Low-dose Long-term Continuous Intravenous Infused 5-fluorouracil Chemotherapy in the Treatment of Stage IV, Recurrent or Metastatic Nasopharyngeal Carcinoma
Brief Title: A Multi-center, Randomized, Double-blind, Phase III Clinical Trial of Leucogen Versus Placebo on Leukocyte and Platelet Whole-course Management Assisted by PFLL Chemotherapy in the Treatment of Stage IV, Recurrent or Metastatic NPC
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: JIANGSU JIBEIER PHARMACEUTICAL CO.,LTD (Unknown)
Responsible Party: Principal Investigator, Yun-fei Xia, Principal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022-FXY-253
Record Dates: First submitted 2023-03-10; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Nasopharyngeal Carcinoma; Leucogen; Chemotherapy; Myelosuppression
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Fluorouracil; lobaplatin; Leyk

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Placebo Comparator): Chemotherapy:
  5-fu: 200mg/m2/d, continuous intravenous infusion on the 1st to 30th day of each cycle; Lobaplatin: 30mg/m2, used on the 1st and 28th day of each cycle; Q60d; Every 2 months for a treatment cycle, use 6 cycles, a total of 12 months.
  Drug: Placebo After diagnosis of stage IV, recurrent or metastatic nasopharyngeal carcinoma (within 3 weeks before treatment), placebo tablets were started,) 2 tablets/dose 3 times for peri-chemotherapy prophylaxis and inter-chemotherapy period, 3 tablets/dose 3 times daily during chemotherapy, and continued to be given orally 2 tablets/dose 3 times daily for 4 weeks after the end of chemotherapy. In case of grade III-IV myelosuppression during treatment, recombinant human granulocyte-stimulating factor injection (manufactured by Qilu Pharmaceutical Co., Ltd.) was given again at 2~5ug/kg, subcutaneously once daily, and the clinical trial was terminated.
  Interventions: Drug: 5-fu; Drug: Lobaplatin; Drug: Placebo
- Experimental group (Active Comparator): Chemotherapy:
  5-fu: 200mg/m2/d, continuous intravenous infusion on the 1st to 30th day of each cycle; Lobaplatin: 30mg/m2, used on the 1st and 28th day of each cycle; Q60d; Every 2 months for a treatment cycle, use 6 cycles, a total of 12 months.
  Drug: Leucogen After the diagnosis of stage IV, recurrent or metastatic nasopharyngeal carcinoma (within 3 weeks before treatment), oral leucogen tablets (manufactured by JIANGSU JIBEIER PHARMACEUTICAL CO.,LTD, 20 mg/tablet) were started and 40 mg/dose was used 3 times for peri-chemotherapy prophylaxis and inter-chemotherapy period, and 60 mg/dose was used 3 times daily during chemotherapy, and 40 mg/dose was continued orally 3 times daily for 4 weeks after the end of chemotherapy. In case of grade III-IV myelosuppression during treatment, recombinant human granulocyte-stimulating factor injection (manufactured by Qilu Pharmaceutical Co., Ltd.) was given again at 2~5ug/kg, subcutaneously once daily, and the clinical trial was terminated.
  Interventions: Drug: 5-fu; Drug: Lobaplatin; Drug: leucogen

INTERVENTIONS:
Drug: 5-fu — 5-fu: 200mg/m2/d, continuous intravenous infusion on the 1st to 30th day of each cycle.
Drug: Lobaplatin — 30mg/m2, used on the 1st and 28th day of each cycle.
Drug: Placebo — 2 tablets/dose 3 times for peri-chemotherapy prophylaxis and inter-chemotherapy period, 3 tablets/dose 3 times daily during chemotherapy, and continued to be given orally 2 tablets/dose 3 times daily for 4 weeks after the end of chemotherapy.
  Arms: Control group
Drug: leucogen — 40 mg/dose was used 3 times for peri-chemotherapy prophylaxis and inter-chemotherapy period, and 60 mg/dose was used 3 times daily during chemotherapy, and 40 mg/dose was continued orally 3 times daily for 4 weeks after the end of chemotherapy.
  Arms: Experimental group

SUMMARY:
Toxic and side effects during and after chemoradiotherapy for nasopharyngeal carcinoma seriously affect patients' treatment compliance and long-term quality of life. Active and effective prediction, prevention and management of toxic and side effects is an important element to improve the prognosis of patients. Leucogen has the ability to promote the growth and maturation of granulocytes in the bone marrow and the proliferation of leukocytes, and is widely used in radiation therapy and chemotherapy-induced leukopenia in malignant carcinomas. In addition, leucogen may have potential anticancer synergistic effects. Therefore, based on the application prospect of leucogen in preventing myelosuppression during chemotherapy for solid tumors, the study was designed to investigate the efficacy and safety of leucogen versus placebo on leukocyte and platelet whole-course management assisted by platinum plus low-dose long-term continuous intravenous infused 5-fluorouracil chemotherapy in the treatment of stage IV, recurrent or metastatic nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old and ≤60 years old；
2. Pathological diagnosis of stage IV, recurrent or distant metastatic nasopharyngeal carcinoma；
3. Patients with stage IV, metastatic (including primary and secondary) or recurrent nasopharyngeal carcinoma who are not suitable for local treatment, local treatment mainly refers to measures related to anti-tumor therapy, including surgery, radiofrequency ablation, transhepatic artery chemoembolization (TACE), radiotherapy (excluding bone metastases, local moderate amount of radiation therapy for symptom relief without affecting hematological indicators)；
4. Karnofsky functional status score should be at least 70 points (the decline of functional status score caused by tumor should be appropriately relaxed after the judgment of the researcher, and the minimum score should be no less than 50 points. );
5. At least 1 measurable lesion according to RECIST1.1 assessment criteria, measurable lesion should not have received local treatment such as radiotherapy;
6. Expected survival ≥3 months;
7. The function of vital organs meets the following requirements (not allowed within 14 days before screening . May use any blood components, cell growth factors, leukoplast, platelets Drugs, anemia correction drugs) :

   * Neutrophil absolute count (ANC) ≥1.5×109/L
   * Platelet ≥100×109/L;
   * Hemoglobin ≥8.0g/ dL (note: Hemoglobin ≥8.0g/ dL can be achieved through blood transfusion or other intervention);
   * Serum albumin ≥2.8g/dL;
   * Bilirubin ≤ 1.5x ULN, ALT and AST≤ 1.5x ULN; ALT and AST≤ 5x ULN if liver metastasis was present;
   * creatinine clearance ≥50mL/min
8. Women of non-surgical sterilization or reproductive age and sexually active men enrolled in the study are required to use a medically effective form of contraception (such as an intrauterine device [IUD], birth control pills or condoms) for the duration of the study treatment and for at least 3 months after the last use of Tamfu and for at least 6 months after the last use of chemotherapy; The serum or urine HCG test of female patients of reproductive age who were not undergoing surgical sterilization must be negative within 7 days prior to study enrollment. And must be non lactation period;
9. Informed consent has been signed. -

Exclusion Criteria:

1. Have a history of allergy to 5-FU, cisplatin and leucogen;
2. Received elevated blood therapy 14 days prior to screening (including cytokines, leuk-lifting drugs, platelet-lifting drugs, anemia-correcting drugs, etc.)
3. Major surgery other than nasopharyngeal cancer was diagnosed within 28 days prior to randomization or major surgery was expected during the study period;
4. The subject has any active autoimmune disease or a history of autoimmune disease (e.g., but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism); Subjects with vitiligo or asthma in complete remission during childhood without any intervention as adults could be included; Subjects with asthma requiring medical intervention with bronchodilators were excluded);
5. Subject is taking immunosuppressants, or systemic, or absorbable sites Hormone therapy to achieve immunosuppression (dose >10mg/ day prednisone or Other equally effective hormones) and continued to be used within 2 weeks prior to enrollment.
6. The subject has previous or co-existing malignancies (except those that have been cured and survived for more than 5 years without cancer, such as basal cell carcinoma of the skin, carcinoma in situ of the cervix and papillary carcinoma of the thyroid);
7. Patients with cardiac clinical symptoms or diseases that are not well controlled, such as: # HEART failure of NYHA grade 2 or above # unstable angina pectoris # myocardial infarction within 1 year # clinically significant ventricular arrhythmias or ventricular arrhythmias requiring treatment or intervention;
8. Subjects have active infection or have unexplained fever >38.5 degrees during screening but before the first dose (the investigator judged that the subjects' fever due to tumor could be included in the study);
9. Subjects with congenital or acquired immune deficiency (e.g. HIV infected), or active hepatitis (reference: HBsAg, anti-HBS, HBeAg, anti-HBC, anti-HBE, HBV DNA≥10#/ml, liver cell transaminase, etc.); Hepatitis C reference: HCV antibodies and HCVRNA);
10. The subject has a known history of psychotropic drug abuse, alcoholism or drug abuse;
11. In the judgment of the researcher, the subject has other factors that may lead to the termination of the study, such as other serious diseases (including mental diseases) requiring combined treatment, serious abnormal laboratory examination, family or social factors, which may affect the safety of the subject, or the collection of test data and samples.
12. Women who are pregnant or breastfeeding, or who refuse/cannot accept medically acceptable conditions. For women with potential pregnancy and sexually active men.

    -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Therapeutic toxicity | Up to 3 approximately months
  Grade I-IV hematological toxicity
Time of myelosuppression | Up to 3 approximately months
  From the beginning of treatment to the onset of myelosuppression

SECONDARY OUTCOMES:
OS | Up to 5 years
  Overall survival
PFS | Up to 5 years
  Progression-free survival
ORR | Up to 2 approximately years
  ORR
DCR | Up to 2 approximately years
  Disease control rate
DOR | Up to 2 approximately years
  Duration of response

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No